CLINICAL TRIAL: NCT01984502
Title: A Phase I CyberKnife Accelerated Hemilarynx Stereotactic Radiotherapy Study for Early-stage Glottic Larynx Cancer
Brief Title: CyberKnife Accelerated Hemilarynx Stereotactic Radiotherapy Study for Early-stage Glottic Larynx Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Baran Sumer, Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 062013-052
Record Dates: First submitted 2013-11-07; First posted 2013-11-14 (Estimated); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Early-stage Glottic Larynx Cancer
Keywords: Larynx Cancer
MeSH Terms: conditions — Laryngeal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Radiation (Experimental): CyberKnife Accelerated Hemilarynx Stereotactic Radiotherapy
  Interventions: Radiation: CyberKnife Accelerated Hemilarynx Stereotactic Radiotherapy

INTERVENTIONS:
Radiation: CyberKnife Accelerated Hemilarynx Stereotactic Radiotherapy — CyberKnife Accelerated Hemilarynx Stereotactic Radiotherapy

SUMMARY:
The feasibility of reducing fractions in early-stage laryngeal cancer has not previously been prospectively studied, and we will therefore conduct a careful phase I bio-equivalent dose fraction reduction study.

DETAILED DESCRIPTION:
Patients enrolled at each dose level will undergo routine evaluations to identify potential toxicities as well functional voice analyses. Adequate waiting periods will be used to ensure that fraction reduction does not proceed prior to observing toxicity. The purpose of the study will be either to determine the maximal fraction reduction possible until a dose is reached where a dose-limiting toxicity occurs. The initial dose and fractionation will be 50 Gy in 15 fractions with the goal to reduce number of fractions to a dose of 42.5 Gy in 5 fractions. The rationale for using 5 fractions is that it is tolerated in centrally located lung tumors at a dose of 50 Gy in 5 fractions, and thus, is likely to be tolerated in large calliber airways.

ELIGIBILITY:
Inclusion Criteria:

3.1.1 Stage Tis, T1, or T2 laryngeal squamous cancer as defined by American Joint Commission on Cancer (AJCC) 2007 staging system

3.1.2 Biopsy proven squamous cell carcinoma histology or squamous cell variants (sarcomatoid, verrucous, basaloid, and papillary subtypes) involving the true vocal cord

3.1.3 Direct laryngoscopy showing no evidence of greater than Stage II true glottic larynx cancer

3.1.4 PET/CT, X-ray, CT-scan of the chest showing no evidence of metastatic disease

3.1.5 PET/CT or CT-scan of the neck showing no evidence of nodal involvement

3.1.6 Age ≥ 18 years.

3.1.7 Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

3.1.7.1 A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

* Has not undergone a hysterectomy or bilateral oophorectomy; or
* Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).

3.1.8 Ability to understand and the willingness to sign a written informed consent

3.1.9 Eastern Cooperative Oncology Group (ECOG) performance status 0-1

3.1.10 Negative Urine β-HCG or negative serum quantitative β-HCG or within 2 weeks prior to registration for women of childbearing potential

Exclusion Criteria:

3.2.1 Evidence of fixed vocal cord (Stage cT3)

3.2.2 Evidence of thyroid or soft tissue invasion (Stage cT4)

3.2.3 Evidence of positive nodal disease (Stage N1)

3.2.4 Evidence of metastatic disease (Stage M1)

3.2.5 Subjects may not be receiving any other investigational agents.

3.2.6 Non-squamous histology including lymphoma, neuroendocrine carcinoma, adenocarcinoma, or other histology.

3.2.7 Previous laryngeal surgery.

3.2.8 Previous laser therapy within one year prior to protocol treatment.

3.2.9 Previous head and neck radiation therapy involving the glottic larynx

3.2.10 Patients with collagen vascular disease, specifically dermatomyositis with a CPK level above normal or active skin rash, systemic lupus erythematosis, or scleroderma.

3.2.11 Any prior treatment with radiation therapy or chemotherapy for the currently diagnosed larynx cancer prior to registration.

3.2.12 History of another active uncontrolled malignancy at the time of study enrollment

3.2.13 Subjects must not be pregnant due to the potential for congenital abnormalities.

3.2.14 Patients smoking in excess of 2 packs of cigarettes per day.

3.2.15 ECOG performance status ≥ 2

3.2.16 Life expectancy < 3 years

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-11-18 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Fraction | 90 days
  To determine the feasibility of fraction reduction for early-stage laryngeal cancer without exceeding the maximum tolerated dose.

SECONDARY OUTCOMES:
overall survival | 5 years
  To determine overall survival at 5 years
loco-regional control | 5 years
  To determine loco-regional control at 5 years as determined by physical exam, visualization of tumor by layngoscopy, and CT-scan of the neck to determine if the primary tumor is controlled. A tissue biopsy or recurrent or persistent disease will be required to be considered a loco-regional failure.
functional voice quality | 18 months
  To characterize functional voice quality of patients treated on this protocol.
Quality of Life | 18 months
  To characterize the HR-QoL and PRO of patients treated on this protocol.
cost-effectiveness | 18 months
  To determine cost-effectiveness of hypofractionated larynx irradiation
late toxicity | 18 months
  To determine late toxicity as defined as treatment-related toxicity occurring ≥ 18 months from completion of radiation therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Baran Sumer, MD, Principal Investigator — UTSW
Locations (1):
- University Of Texas Southwestern Medical Center, Dallas, Texas, United States

REFERENCES:
- [Derived] Zhang Y, Chiu T, Dubas J, Tian Z, Lee P, Gu X, Yan Y, Sher D, Timmerman R, Zhao B. Benchmarking techniques for stereotactic body radiotherapy for early-stage glottic laryngeal cancer: LINAC-based non-coplanar VMAT vs. Cyberknife planning. Radiat Oncol. 2019 Nov 4;14(1):193. doi: 10.1186/s13014-019-1404-z. PMID 31684993
- [Derived] Schwartz DL, Sosa A, Chun SG, Ding C, Xie XJ, Nedzi LA, Timmerman RD, Sumer BD. SBRT for early-stage glottic larynx cancer-Initial clinical outcomes from a phase I clinical trial. PLoS One. 2017 Mar 2;12(3):e0172055. doi: 10.1371/journal.pone.0172055. eCollection 2017. PMID 28253270